CLINICAL TRIAL: NCT06600711
Title: Randomized Control Trial of Nitazoxanide for the Treatment of Cryptosporidium Infection in Malnourished Children in Bangladesh
Brief Title: Nitazoxanide for Treatment of Cryptosporidium in Children
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Johns Hopkins Bloomberg School of Public Health (Other)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IRB00024940; U01AI167788-01A1 (NIH)
Record Dates: First submitted 2024-09-16; First posted 2024-09-19 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Cryptosporidiosis
Keywords: Nitazoxanide
MeSH Terms: conditions — Cryptosporidiosis | interventions — nitazoxanide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Nitazoxanide (Experimental)
  Interventions: Drug: Nitazoxanide
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Nitazoxanide — 5 mL suspension (100 mg), 2x/day for 3 days
  Arms: Nitazoxanide
Drug: Placebo — identical in consistency, appearance, and taste to nitazoxanide suspension. 5 mL suspension given 2x/day for 3 days
  Arms: Placebo

SUMMARY:
The goal of this clinical trial is to learn if nitazoxanide (NTZ) can treat Cryptosporidium infection in children age 6-12 months. The main questions it aims to answer are:

* Does NTZ treatment of diarrheal Cryptosporidium infection lower the number of days of diarrhea?
* Does NTZ treatment of diarrheal and non-diarrheal Cryptosporidium infection lower the number of days that parasites can be found in the stool?

Researchers will compare NTZ to a placebo (a look-alike substance that contains no drug) to see if NTZ works to treat Cryptosporidium.

Participants will:

* Take NTZ or placebo for 3 days
* Receive regular visits from field research assistants
* Provide blood and urine samples

ELIGIBILITY:
Inclusion Criteria:

* tests positive for Cryptosporidium by stool point-of-care test, with or without active diarrhea
* family plans on remaining in the area for next 6 months

Exclusion Criteria:

* history of hypersensitivity to nitazoxanide.
* taking warfarin. Tizoxanide, the metabolite of nitazoxanide is highly bound to plasma proteins and may compete with binding sites of other highly plasma bound drugs with narrow therapeutic indices, including warfarin.
* history of renal insufficiency or a baseline serum creatinine = 40 µmol/L. Renal clearance of the drug has not been studied.
* history of hepatic dysfunction or serum aspartate aminotransferase (AST) ;
* 50 U/L, serum alanine transaminase (ATL) ;
* 50 U/L, or serum bilirubin ;
* 23 µmol/L. Hepatic clearance of the drug has not been studied.

Ages: 6 Months to 12 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 480 (Estimated)
Dates: Start 2026-04-01 (Estimated); Primary Completion 2028-12 (Estimated); Study Completion 2030-05 (Estimated)

PRIMARY OUTCOMES:
Days of Cryptosporidium-associated diarrhea | 7 days
Time to clearance of Cryptosporidium from stool | 6 months
  Measured in days

SECONDARY OUTCOMES:
Adverse events, total and stratified by age | 6 months
Time-to-first Cryptosporidium infection in sibling | 6 months
  Measured in days
Change in weight from baseline to 6 months post-treatment | Baseline, 6 months
  Weight measured in kilograms
Change in Lactulose:Mannitol ratio from baseline to 6 months post treatment | Baseline, 6 months
Change in height-for-age adjusted z-score from baseline to 6 months post treatment | Baseline, 6 months
  Measured in centimeters

CONTACTS AND LOCATIONS:
Overall Officials: Poonum Korpe, MD, Principal Investigator — Johns Hopkins University